CLINICAL TRIAL: NCT04899427
Title: Orelabrutinib Combined With PD-1 Inhibitor in Relapsed/Refractory Primary Central Nervous System Lymphoma: a Prospective Multi-center Phase II Study
Brief Title: Phase II Study of Orelabrutinib Combined With PD-1 Inhibitor in Relapsed/Refractory Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Beijing Tongren Hospital (Other); Beijing Luhe Hospital (Other); Shanxi Province Renmin Hospital (Unknown); Henan Cancer Hospital (Other Government); Henan Province Renmin Hospital (Unknown); The Second Affiliated Hospital of Dalian Medical University (Other); Hebei Medical University Fourth Hospital (Other); The First Hospital of Chinese Medical University (Unknown); Qilu Hospital of Shandong University (Other); The First Hospital of Zhengzhou University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-009
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Primary Central Nervous System Lymphoma; orelabrutinib; PD-1 inhibitor; Overall response rate
MeSH Terms: interventions — orelabrutinib; sintilimab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orelabrutinib combined with PD-1 inhibitor (Experimental): The experimental arm will be treated orelabrutinib plus PD-1(programmed death）inhibitor every 21 days as one cycle. The responses will be evaluated every 2 cycles during the first 6 cycles and every 3 months until progression.
  The investigators can choose Sintilimab Injection or Tislelizumab Injection at the beginning of treatment，but they can't exchange to another during the whole treatment.
  Interventions: Drug: orelabrutinib; Drug: Sintilimab; Drug: Tislelizumab

INTERVENTIONS:
Drug: orelabrutinib — Orelabrutinib will be given as 150mg per day orally, until progression of the disease (PD), unacceptable toxicity, or patient/investigator discretion.
Drug: Sintilimab — Sintilimab 200mg intravenous infusion d1, every 21 days for 1 cycle. The medicine will be given until progression of the disease (PD), unacceptable toxicity, or patient/investigator discretion.
Drug: Tislelizumab — Tislelizumab 200mg intravenous infusion d1, every 21 days for 1 cycle. The medicine will be given until progression of the disease (PD), unacceptable toxicity, or patient/investigator discretion.

SUMMARY:
This is a prospective multicenter single-arm phase II study, and the purpose of this study is to evaluate the efficiency of Orelabrutinib combined with PD-1 inhibitor regimen relapsed/refractory primary intraocular lymphoma. Overall response rate （ORR） after 4 cycles is the primary endpoint.

DETAILED DESCRIPTION:
All the patients will be treated with Orelabrutinib combined with PD-1 inhibitor ：Orelabrutinib 150mg qd，Tislelizumab Injection 200mg d1 or Sintilimab injection 200mg d1， every 21-day for 1 cycle). Patients will be evaluated every 2 cycles by MRI scan during the first 6 cycles，and then the interval of investigation will be prolonged to 12 weeks. The patients who achieved complete remission (CR) or partial remission (PR) or stable disease (SD) will receive further treatment. The patients progressed disease (PD) will withdraw from the trial and receive salvage regimens. The treatment will be continued for 2 years or until progression of the disease (PD), unacceptable toxicity, or patient/investigator discretion.

During following-up, surveillance ophthalmologic examination and brain magnetic resonance imaging (MRI) scans can be performed every 3 months up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old ≤75 Years old, male or female
* Primary Central nerves system lymphoma confirmed by cytology or histology according to WHO2016 criteria
* No evidence of systemic lymphoma
* Patients with a clear diagnosis of relapsed and/or refractory PCNSL: they received at least one regimen containing methotrexate.
* At least one measurable lesion according to Lugano 2014 criteria
* Adequate organ function and adequate bone marrow reserve

Exclusion Criteria:

* Malignant tumors other than B-NHL within 5 years prior to screening, except cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and breast ductal carcinoma in situ after radical surgery
* Active HIV, HBV, HCV or treponema pallidum infection
* Any instability of systemic disease, including but not limited to active infection (except local infection), severe cardiac, liver, kidney, or metabolic disease need therapy
* Female subjects who have been pregnant or breastfeeding, or who plan to conceive during or within 1 year after treatment, or male subjects' partner plans to conceive within 1 year after their cell transfusion
* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment
* Any systemic antitumor therapy performed within 2 weeks before enrollment
* Previous use of other BTK inhibitors or PD-1 inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-03-24 (Estimated); Study Completion 2023-10-24 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 3 weeks after the end of 4 cycles of induction (each cycle is 21 days)
  ORR was calculated by the proportion of patients who achieved complete remission and partial remission.

SECONDARY OUTCOMES:
1 years progression-free survival | from the date of treatment to the subject finished his 1 years follow-up phase or the disease relapsed or the death due to lymphoma
  1 years progression-free survival was calculated from the date of therapy until death from lymphoma or 1-year follow up without relapsing

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Zhang, Beijing, Beijing Municipality, China